CLINICAL TRIAL: NCT00975273
Title: Targeting CO2 Levels in Breathing Training for Asthma
Brief Title: Breathing Training for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Baylor Health Care System (Other)
Responsible Party: Principal Investigator, Alicia Meuret, Associate Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01HL89761-2; SMU IRB:KS08-051; Baylor IRB: 001-180; 5R01HL089761 (NIH)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: ASTHMA
Keywords: Asthma; Dyspnea; Paroxysmal; Pulmonary; Respiratory hypersensitivity; Airway inflammation; Airway obstruction; Wheezing
MeSH Terms: conditions — Asthma; Dyspnea; Respiratory Hypersensitivity; Airway Obstruction; Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breathing Training (Experimental): Patients will receive biofeedback assisted breathing training
  Interventions: Behavioral: Capnometry Assisted Respiration Training
- Breathing Awareness (Active Comparator): Patients will receive biofeedback assisted breathing awareness training.
  Interventions: Behavioral: Breathing Awareness

INTERVENTIONS:
Behavioral: Capnometry Assisted Respiration Training — Patients learn to alter their breathing pattern by breathing abdominally, slowly, regularly, and shallowly in order to raise their PCO2 levels with the assistance of a biofeedback device.
  Other Names: CART
  Arms: Breathing Training
Behavioral: Breathing Awareness — Patients learn to alter their breathing pattern by breathing abdominally, slowly, regularly using a biofeedback device.
  Arms: Breathing Awareness

SUMMARY:
For the proposed randomized controlled treatment study, the investigators plan to compare the effects of this hypoventilation-based breathing training with a control intervention that will focus on breathing regularity and awareness. The two therapeutic procedures are closely matched on important variables such as duration and the nature of patient-therapist interaction, monitoring asthma related status and the medication intake, use of scientific equipment and monitoring devices to increase adherence, and initial plausibility. Asthma patients who will be evaluated before, during, directly after, and at 2 months and 6 months after training.

DETAILED DESCRIPTION:
For this randomized controlled treatment study, the investigators plan to compare the effects of hypoventilation-based breathing training with a control intervention that will focus on breathing regularity and awareness. The two therapeutic procedures are closely matched on important variables such as duration and the nature of patient-therapist interaction, monitoring asthma related status and the medication intake, use of scientific equipment and monitoring devices to increase adherence, and initial plausibility. Asthma patients will be evaluated before, during, directly after, and at 1 month and 6 months after training. The primary goal of this training is to determine if a capnometry-assisted breathing training to raise end-tidal CO2 will produce more improvement in asthma control than a control training of breathing awareness. The second goal is to determine if capnometry-assisted breathing training for raising pCO2 will lead to higher pCO2 levels after training than before training on all three measures of pCO2 (the 2-hour monitoring, the standardized training sessions, and the homework assignments). The last objective is to determine if the clinical improvement in asthma outcomes for the raise-pCO2 breathing group will be greater in patients with more improvement in their pCO2.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 18 and 65 years of age
2. Understand and read english adequately
3. A previously documented history of asthma from intermittent to severe (symptoms plus objective documentation of at least partially reversible airflow obstruction)
4. Willing to undergo a 5-session course of breathing training
5. Current asthma symptoms

Exclusion Criteria:

1. Clinically significant heart disease
2. Clinically significant cerebrovascular disease
3. Clinically significant thyroid dysfunction
4. Out-of-control diabetes
5. Use of oral corticosteroids in the last 3 months
6. Active smokers or more than 10 pack years
7. Clinically significant chronic obstructive pulmonary disease
8. Clinically significant emphysema
9. Current alcohol and substance dependence
10. Psychotic disorders and high risk for personality disorders
11. Having received previous breathing training exercises for asthma
12. Not willing to abstain from taking the morning dose of their long-term bronchodilator or leukotriene inhibitors or from using their short-acting beta-2 adrenergic agonists or anticholinergic bronchodilators for 8 hours before the pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up assessments (Medication withdrawal will be discouraged if patients should experience significant symptoms before the assessments. They will be offered to reschedule the appointment without any consequences for their enrollment in the study.)
13. Night shift workers
14. Tuberculosis
15. Pregnant, plan on becoming pregnant, or nursing during the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
pCO2 levels (as an indicator of training manipulation success) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions, patients perform self-assessments on a daily basis throughout, pre- and post-treatment 2h monitoring
diurnal PEF variability (as an indicator of asthma pathophysiology and control) | pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up
Asthma Control Test (as a self-report indicator of asthma control) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up. Further assessments will be made at the beginning of each of the five weekly training sessions.

SECONDARY OUTCOMES:
respiration rate from capnometry and further measures of ventilation from ambulatory recordings (as further indicators of training manipulation success) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions, patients perform self-assessments on a daily basis throughout, pre- and post-treatment 2h monitoring
FeNO | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions
airway hyperreactivity by methacholine | at pretreatment and optionally at 1 month follow up
spirometric lung function and respiratory resistance (as further indicators of asthma pathophysiology) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions, patients perform self-assessments on a daily basis throughout.
reported symptoms | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions, patients perform self-assessments on a daily basis throughout
monitored bronchodilator use | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions, patients record usage throughout treatment
reported inhaled corticosteroid use (as self-report and behavioral indicators of asthma control) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions
effects on perceived general control of asthma management, asthma self-efficacy, and impact and control of asthma triggers (as an indicator of asthma self-management) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions
physical and mental health status, stress, anxiety and depression (as indicators of general well-being) | Measured at pre-treatment, post-treatment, 1-month follow-up, and 6-month follow-up, at the beginning of each of the five weekly training sessions

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Meuret, PhD, Principal Investigator — SMU; Thomas Ritz, PhD, Principal Investigator — SMU; Mark Millard, MD, Principal Investigator — BUMC
Locations (2):
- United States (2):
  - Baylor University Medical Center (BUMC), Dallas, Texas
  - Southern Methodist University (SMU), Dallas, Texas

REFERENCES:
- [Derived] Meuret AE, Rosenfield D, Millard MM, Ritz T. Biofeedback Training to Increase P co2 in Asthma With Elevated Anxiety: A One-Stop Treatment of Both Conditions? Psychosom Med. 2023 Jun 1;85(5):440-448. doi: 10.1097/PSY.0000000000001188. Epub 2023 Mar 23. PMID 36961348
- [Derived] Ritz T, Rosenfield D, Steele AM, Millard MW, Meuret AE. Controlling asthma by training of Capnometry-Assisted Hypoventilation (CATCH) vs slow breathing: a randomized controlled trial. Chest. 2014 Nov;146(5):1237-1247. doi: 10.1378/chest.14-0665. PMID 25122497